CLINICAL TRIAL: NCT00272545
Title: Adaptation of a CBT Intervention for Eating Disorders
Brief Title: Effectiveness of a Normalization of Eating Intervention Program for Treating Women With Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH071691 (NIH); R34MH071691 (NIH); DATR A2-AIR
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Eating Disorders
Keywords: Anorexia Nervosa; Bulimia Nervosa; Cognitive Behavioral Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa | interventions — Therapeutics

ARMS (2):
- 1 (Experimental): Participants will receive the normalization of eating program
  Interventions: Behavioral: Normalization of Eating (NOE)
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Normalization of Eating (NOE) — The NOE is a 6-week program based on principles of CBT. Participants will receive individual therapy, as well as take part in group and family therapy sessions. In addition, participants will be supervised while eating meals.
  Arms: 1
Behavioral: Treatment As Usual (TAU) — Treatment as usual will include standard care for a person with an eating disorder.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a new approach to a normalization of eating program, based on principles of cognitive-behavioral therapy, in treating women with anorexia nervosa or bulimia nervosa.

DETAILED DESCRIPTION:
Eating disorders are real, treatable medical illnesses. They are often characterized by disturbances in eating behavior, such as drastic reduction of food intake or extreme overeating, as well as feelings of distress or extreme concern about body shape or weight. The two main types of eating disorders are anorexia nervosa and bulimia nervosa. A third type, binge-eating disorder, is pending approval as a formal psychiatric diagnosis. Eating disorders frequently develop during adolescence or early adulthood, and they occur more often in females than in males. Studies have shown cognitive behavioral therapy (CBT) to be the most effective approach to treating eating disorders. However, the applicability of these findings to clinical settings and intensive outpatient therapy programs (IOPs) remains unknown. This study will evaluate the effectiveness of a new approach to a normalization of eating (NOE) program, based on principles of CBT, in treating women with anorexia nervosa or bulimia nervosa.

Participants in this open-label study will be assigned to receive either treatment-as-usual (TAU) or NOE. Participants admitted to the study in the first 8 months of the trial will receive TAU. Those admitted after the first 8 months will take part in the NOE program. Participants may begin receiving treatment as soon as they enter the study and will continue receiving their assigned treatments for 6 weeks. All participants in the NOE group will be required to report to the study site three evenings a week. They will receive individual therapy, as well as take part in group and family therapy sessions. In addition, they will be supervised while eating a meal. Body weight, results of the Eating Disorders Examination and the Structured Clinical Interview for DSM-IV Axis I disorders, and self-report measures will be assessed post-treatment and at the Month 6 follow-up visit.

Note: Participants are recruited from the Renfrew Center's outpatient programs located in the Philadelphia area. Individuals outside of Renfrew cannot volunteer for this study. For more information about the Renfrew Center's inpatient or outpatient treatment programs, please call 1-800-RENFREW.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an eating disorder or eating disorder not otherwise specified (except for binge eating disorder), as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association
* Agrees to remain in IOP treatment for at least 3 weeks
* Seeking treatment in one of the Renfrew Center's outpatient programs located in the Philadelphia area

Exclusion Criteria:

* Diagnosis of eating disorder not otherwise specified, including binge eating disorder
* Diagnosis of a psychotic disorder
* Transferred to inpatient treatment during the IOP stay because of worsening health

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Body weight | Measured at baseline, discharge, and 6 month follow-up
Structured Clinical Interview | Measured at baseline
Self-report | Measured at baseline, discharge, and 6 month follow-up
Eating Disorders Examination | Measured at baseline, discharge, and 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Lowe, PhD, Principal Investigator — Drexel University
Locations (1):
- The Renfrew Center of Radnor, Radnor, Pennsylvania, United States